CLINICAL TRIAL: NCT01387009
Title: Acquisition of Normative Data for Musculoskeletal Ultrasound in Children
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Johannes Roth, MD, Children's Hospital of Eastern Ontario
Other Study IDs: IMM 10-0049
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Normative Data Study of Joints of Healthy Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
The primary objective is to establish normative data for Canadian children for the shoulder, elbow, wrist, finger, hip, knee, ankle and toe joint including the relevant tendons surrounding the joint.

DETAILED DESCRIPTION:
The respective joints will be assessed through ultrasonography and data will be collected and analyzed

ELIGIBILITY:
Inclusion Criteria:

* Healthy children

Exclusion Criteria:

* Do not suffer from any condition that might have an effect on their joints.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy children will be recruited via invitation by investigators
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Roth, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Johannes Roth, Ottawa, Ontario, Canada